CLINICAL TRIAL: NCT03240393
Title: Phase II Multicenter 3-cohort Study of Oral cMET Inhibitor INC280 in Chinese Patients With EGFR Wild-type Advanced Non-small Cell Lung Cancer (NSCLC) Who Have Received 1 or 2 Prior Lines of Systemic Therapy for Advanced/Metastatic Disease
Brief Title: Study of Oral cMET Inhibitor INC280 in Chinese Patients With EGFR Wild-type Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280A2202
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma; Non-Small-Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; NSCLC; INC280; EGFR wild-type (wt); advanced non-small cell lung cancer; advanced/metastatic disease; Non-small cell lung carcinoma (NSCLC); treatment of lung cancer after first metastasis; lung cancer; lung adenocarcinoma; Non small cell lung carcinoma; Non-small cell lung cancer; MET exon 14 deletion; MET exon 14 skipping; MET exon 14 mutation; MET mutation; MET amplification; MET inhibitor; MET dysregulation; MET activation; MET signaling; MET pathway; MET; cMET
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms; Adenocarcinoma of Lung | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cMET GCN ≥ 6 (Experimental): Pre-treated patients with cMET GCN ≥ 6 treated with INC280 at 400mg BID
  Interventions: Drug: INC280
- cMET GCN ≥ 4 and < 6 (Experimental): Pre-treated patients with cMET GCN ≥ 4 and < 6 treated with INC280 at 400 mgBID
  Interventions: Drug: INC280
- cMET mutations (Experimental): Pre-treated patients with cMET mutations regardless of cMET GCN treated with INC280 at 400mg BID
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: INC280 — cMET GCN ≥ 6 cMET GCN ≥ 4 and < 6 cMET mutations
  Other Names: capmatinib

SUMMARY:
A phase II study to evaluate antitumor activity of oral cMET inhibitor INC280 in adult Chinese patients with EGFR wild-type, advanced non-small cell lung cancer (NSCLC) who have received one or two prior lines of systemic therapy for advanced/metastatic disease as measured by overall response rate (ORR). The study will also evaluate safety and pharmacokinetics of INC280.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB or IV NSCLC (any histology) at the time of study entry
* Histologically or cytologically confirmed diagnosis of NSCLC that is:

  1. EGFR wt as per patient standard of care by a validated test
  2. AND ALK-negative rearrangement as part of the patient standard of care by a validated test
  3. AND (by central assessment) either:

     * Cohort 1: Pre-treated patients with cMET GCN ≥ 6 or
     * Cohort 2: Pre-treated patients with cMET GCN ≥4 and < 6, or
     * Cohort 3: Pre-treated patients with cMET mutations regardless of cMET GCN, or
* Patients must have failed one or two prior lines of systemic therapy for advanced/metastatic disease
* At least one measurable lesion as defined by RECIST 1.1
* Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1 (CTCAE v 4.03). Patients with any grade of alopecia are allowed to enter the study.
* Patients must have adequate organ function
* ECOG performance status (PS) of 0 or 1

Details and other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Prior treatment with crizotinib, or any other cMET or HGF inhibitor
* Patients with characterized EGFR mutations that predict sensitivity to EGFR therapy, including, but not limited to exon 19 deletions and exon 21 mutations
* Patients with characterized ALK-positive rearrangement
* Clinically significant, uncontrolled heart diseases.
* Patients receiving treatment with medications that cannot be discontinued at least 1 week prior to first INC280 treatment and for the duration of the study:

  * Strong and moderate inhibitors of CYP3A4
  * Strong inducers of CYP3A4
* Impairment of GI function or GI disease that may significantly alter the absorption of INC280
* Patients receiving treatment with any enzyme-inducing anticonvulsant
* Previous anti-cancer and investigational agents within 4 weeks or ≤ 5 x half-life of the agent (whichever is longer) before first dose
* Pregnant or nursing women
* Women of child-bearing potential, unless they are using highly effective methods of contraception
* Sexually active males unless they use a condom during intercourse

Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-31 (Estimated); Primary Completion 2021-10-26 (Estimated); Study Completion 2021-10-26 (Estimated)

PRIMARY OUTCOMES:
ORR based on Central Radiology review/assessment (BIRC) | at least 18 weeks
  Proportion of patients with a best overall response defined as complete response (CR) or partial response (PR) by Blinded Independent Review Committee (BIRC) assessment per RECIST 1.1

SECONDARY OUTCOMES:
Duration of Response (DOR) by BIRC - Key Secondary | at least 18 weeks
  Calculated as the time from the date of the first documented CR or PR by Blinded Independent Review Committee (BIRC) per RECIST 1.1 to the first documented progression or death due to any cause for patients with PR or CR.
ORR by Investigator | at least 18 weeks
  ORR (complete response (CR)+ partial response (PR)) per RECIST 1.1 by investigator assessment
Duration of Response (DOR) by investigator | at least 18 weeks
  DOR per RECIST 1.1 by investigator assessment
Time to Response (TTR) by BIRC | at least 18 weeks
  TTR per RECIST 1.1 by BIRC assessment
Time to Response (TTR) by investigator | at least 18 weeks
  TTR per RECIST 1.1 by investigator assessment
Disease Control Rate (DCR) by BIRC | at least 18 weeks
  DCR per RECIST 1.1 by BIRC assessment
Disease Control Rate (DCR) by investigator | at least 18 weeks
  DCR per RECIST 1.1 by investigator assessment
Progression-free Survival (PFS) by BIRC | at least 18 weeks
  PFS per RECIST 1.1 by BIRC assessment
Progression-free Survival (PFS) by investigator | at least 18 weeks
  PFS per RECIST 1.1 by investigator assessment
Overall Survival (OS) | at least 18 weeks
  OS, defined as time from first dose of INC280 to death due to any cause
Cmax profile of INC280 | 6 weeks
  Pharmacokinetics of INC280
Cmax profile of INC280 metabolite CMN288 | 6 weeks
  Pharmacokinetics of INC280 metabolite CMN288
Cmin profile of INC280 | 6 weeks
  Pharmacokinetics of INC280
Cmin profile of INC280 metabolite CMN288 | 6 weeks
  Pharmacokinetics of INC280 metabolite CMN288
Plasma concentration-time profiles of INC280 | 6 weeks
  Pharmacokinetics of INC280
Plasma concentration-time profiles of INC280 metabolite CMN288 | 6 weeks
  Pharmacokinetics of INC280 metabolite CMN288

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided
Planned Shared Data Description: Copy and paste this Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com